CLINICAL TRIAL: NCT04090931
Title: A Clinical Comparison of the Effectiveness of Two Types of Orthodontic Aligning Archwire Materials: A Randomized Clinical Trial
Brief Title: A Clinical Comparison of the Effectiveness of Two Types of Orthodontic Aligning Archwire Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Yassir A. Yassir, Assistant Professor of Orthodontics, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of Baghdad
Record Dates: First submitted 2019-09-09; First posted 2019-09-16 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Teeth; Anomaly, Position
MeSH Terms: conditions — Congenital Abnormalities | interventions — Orthodontics

STUDY DESIGN:
Intervention Model Description: Orthodontic patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding to treatment allocation was possible only for the investigator and data analyst because the clinicians could know the type of archwiers from their flexibility. All the trial documents were labeled with the study ID number, which was used for participant identification and data collection without unmasking the allocation group. This allowed the investigator to complete data collection and measurements blindly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-Activated Nickel-Titanium Archwires (Experimental): Heat-activated NiTi (HANT) Group (TruFlex™ Thermal Nickel-Titanium, Ortho Technology, USA):
  * 0.014-inch HANT
  * 0.016-inch HANT
  Interventions: Procedure: Orthodontic treatment
- Superelastic Nickel-Titanium Archwires (Experimental): Superelastic NiTi (SENT) Group (TruFlex™ Nickel-Titanium, Ortho Technology, USA):
  * 0.014-inch SENT
  * 0.016-inch SENT
  Interventions: Procedure: Orthodontic treatment

INTERVENTIONS:
Procedure: Orthodontic treatment — leveling and aligning stage in orthodontics

SUMMARY:
The aim of this study is to compare the effectiveness of using heat-activated NiTi with superelastic NiTi archwires during the initial phase of orthodontic treatment.

Primary Objective:

To compare the difference in the amount of crowding in the lower incisors after 4 and 8 weeks from the start of treatment.

Secondary Objectives:

1. To compare the amount of orthodontically-induced inflammatory root resorption (OIIRR) in the apical region of mandibular central incisors between the two groups of archwires
2. To compare the amount of pain perception between the two groups of archwires during the 1st week after each wire placement.

DETAILED DESCRIPTION:
Objectives: To compare the heat-activated nickel titanium (HANT) with superelastic nickel titanium (SENT) archwires in terms of their effectiveness in aligning teeth, possibility of inducing root resorption, and patient perception of pain during the initial phase of treatment.

Subjects and Methods: Orthodontic patient aged 12 years or over with lower anterior crowding of 3-6 mm. who need treatment without extraction, were randomly allocated to the HANT and SENT archwires groups with a 1:1 allocation ratio. Archwire sequence in both groups was 0.014-inch and 0.016-inch, respectively. Each archwire was placed for 4 weeks. Outcome measures included the amount of crowding using Little's irregularity index (LII), apical root resorption, and pain perception. The effectiveness of alignment was tested using 2X2 mixed factorial ANOVA, while root resorption and pain perception were tested by the Mann-Whitney U test, and Wilcoxon signed-rank test (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for fixed appliance orthodontic treatment who have a moderate crowding (3-6mm) according to the Little's irregularity index (LII).
2. Full set of lower permanent dentition excluding the third molars.
3. No history of trauma or root resorption in the lower incisors.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Less than 3mm of lower incisor crowding (LII) or with spaced incisors.
3. Severe crowding in the lower arch (greater than 7mm) which requires extraction.
4. Blocked-out teeth that cannot be engaged with the aligning archwire.
5. Patients with periodontally compromised teeth.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome (Alignment efficiency) | 2 months
  The study models, which should be free from any inconsistency (such as bubbles), were used to measure the Little's irregularity index (Little, 1975). This was calculated using a digital Vernier caliper to measure the extent of mesial and distal contact displacement from the mesial contact point of lower canine to that on the other side (to the nearest 0.01mm).

SECONDARY OUTCOMES:
Root resorption | 2 months
  Root resorption was evaluated pre-treatment and after 8 weeks using periapical X-ray with digital X-ray sensors (ATECO). Radiographic films were positioned using a customized sensor holder for the lower anterior teeth with a 7cm film-cone distance using long cone paralleling technique. The radiographs were made at 70kV and 8mA DC with an exposure of 0.25 seconds.
Pain perception | 2 months
  Evaluations of pain/discomfort was made in the evening on a daily basis over the first 7 days after bonding using a 10-point visual analog scale (VAS) of 10cm length. The highest pain level experienced should be reported by each patient. The recording sheet was received by all the patients on the day of bonding, it included seven visual analog scales (one for each day) and the patients were given oral instructions on how to finish the VAS by marking the point on the line which supposed to represent the maximum pain that they felt per day, with 0 refers to "no pain" and 10 refers to "intolerable pain". Patients were reminded daily by a phone call or a text message to mark the recording sheet and to bring it on their next appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- Yassir A. Yassir, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Materials, Methods, Results

REFERENCES:
- [Derived] Nabbat SA, Yassir YA. A clinical comparison of the effectiveness of two types of orthodontic aligning archwire materials: a multicentre randomized clinical trial. Eur J Orthod. 2020 Dec 2;42(6):626-634. doi: 10.1093/ejo/cjz102. PMID 32011678